CLINICAL TRIAL: NCT00620087
Title: Evaluation of a Small Field of View Gamma Camera for Scintimammography in Patients With Atypical Ductal Hyperplasia, Atypical Lobular Hyperplasia, and Lobular Carcinoma In Situ
Brief Title: Molecular Breast Imaging in Women With Atypia and LCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Deborah Rhodes, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1204-03; KG090823 (Other: Susan G. Komen for the Cure); UL1TR000135 (NIH); NCT00963014 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-02-21 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Atypical Lobular Hyperplasia; Atypical Ductal Hyperplasia; Lobular Carcinoma in Situ
Keywords: Atypical lobular hyperplasia; Atypical ductal hyperplasia; Lobular carcinoma in situ; Molecular Breast Imaging
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diagnostic Arm (Other): Women with core-biopsy proven atypia, LCIS, or radial scar who have not yet undergone surgical excision were enrolled in the diagnostic arm. A molecular breast imaging study will be obtained.
  Interventions: Procedure: Molecular Breast Imaging
- Surveillance arm (Other): Women with a diagnosis of ADH, ALH, or LCIS within the past 5 years were enrolled in the surveillance arm. A molecular breast imaging study was done at enrollment (Year 0) and repeated at Yer 2 and Year 4. Patients continued with routine screening mammography during this time period.
  Interventions: Procedure: Molecular Breast Imaging; Procedure: Screening Mammography

INTERVENTIONS:
Procedure: Molecular Breast Imaging — Molecular breast Imaging is a new nuclear medicine technique for imaging the breast. It uses small filed of view semiconductor-based gamma cameras that use Cadmium Zinc Telluride detectors. These have superior spatial and energy resolution to conventional sodium iodide detectors.
Procedure: Screening Mammography — A screening mammogram is used to look for signs of breast cancer in women who don't have any breast symptoms or problems. X-ray pictures of each breast are taken from 2 different angles.
  Arms: Surveillance arm

SUMMARY:
We aim to determine if Molecular Breast Imaging (a new nuclear medicine technique developed at Mayo) can identify malignant breast lesions in women who have atypical ductal hyperplasia, atypical lobular hyperplasia, or lobular carcinoma in situ.

DETAILED DESCRIPTION:
Management of atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH), and lobular carcinoma in situ (LCIS) diagnosed by breast needle core needle biopsy is controversial. Current practice is to recommend excisional biopsy to rule out malignant lesions, which have been reported in more than half of cases in some series. No consistent clinical, pathologic, or radiologic factors have been identified to select patients who do not require surgical excision. This is due, in part, to overlap in the mammographic features of benign and malignant lesions. Furthermore, reliance on mammography for surveillance of these high-risk patients is problematic. This highlights the need for a complementary imaging modality to improve the radiologic distinction between benign and malignant tumors and improve post-biopsy surveillance.

We are evaluating a new semiconductor-based gamma camera which we call Molecular Breast Imaging (MBI) which improves resolution by a factor of 2-3 compared to conventional gamma cameras, and, unlike mammography, is not affected by breast density. Preliminary clinical studies (IRB 0-1761-01)) have shown that scintimammography (SM) using Tc-99m sestamibi and the CZT camera (CZT-SM) has a high sensitivity and specificity for the evaluation of small (5-10 mm) lesions seen on mammography. We hypothesize that the MBI will reliably distinguish lesions that require excisional biopsy from lesions that do not. A secondary aim is to compare the role of MBI with mammography in post-biopsy surveillance.

We aim to enroll 50 Mayo patients who have received a diagnosis of ADH, ALH, or LCIS on core biopsy, who have not yet undergone excisional biopsy, and who consent to undergo MBI of both breasts. For images in which there is discordance with mammographic findings, ultrasound will be used to determine if additional abnormalities warrant excision. Using pathologic correlation, we will determine: 1) If residual foci of ADH, ALH, and LCIS are visible on MBI images; and 2) If MBI images can reliably predict contiguous or separate foci of malignant lesions in either breast.

ELIGIBILITY:
Inclusion Criteria for Surveillance Arm:

* Diagnosis of biopsy-prove ADH, ALH, or LCIS within the past 5 years based on core needle biopsy and/or excisional biopsy and confirmed by a Mayo pathologist.

Inclusion Criteria for Diagnostic Arm:

* Recent core needle biopsy of the breast demonstrating ADH, ALH, or LCIS confirmed by Mayo pathologist.

Exclusion Criteria:

* They are unable to understand and sign the consent form
* They are pregnant or lactating
* They are physically unable to sit upright and still for 40 minutes
* They are younger than 18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Correlation between molecular breast imaging findings and surgical pathology | five years

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J. Rhodes, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rhodes DJ, Hruska CB, Conners AL, Tortorelli CL, Maxwell RW, Jones KN, Toledano AY, O'Connor MK. Journal club: molecular breast imaging at reduced radiation dose for supplemental screening in mammographically dense breasts. AJR Am J Roentgenol. 2015 Feb;204(2):241-51. doi: 10.2214/AJR.14.13357. PMID 25615744